CLINICAL TRIAL: NCT03886987
Title: Skin Sensitization Test (Modified Draize-95 Test) to Support a Low Dermatitis Potential Claim
Brief Title: Skin Sensitization Test (Modified Draize-95 Test)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Medicare Sdn. Bhd. (Industry)
Collaborators: Consumer Product Testing Company, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CTYP01-001
Record Dates: First submitted 2019-03-18; First posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Skin Sensitisation
Keywords: Modified Draize-95 Test; Skin Sensitisation; Repeat Insult Patch Test

STUDY DESIGN:
Intervention Model Description: Blue Non Sterile Powder Free Nitrile Examination Gloves Dose: Approximately 2cm x 2cm square positioned to ensure that the inside portion of the test material maintained skin contact.
  Positive control: 0.4% sodium lauryl sulfate (SLS) Dose: 0.2 ml
  Negative control: Blank patch Dose: Not applicable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Device and Control (Experimental): Blue Non Sterile Powder Free Nitrile Examination Gloves Dose: Approximately 2cm x 2cm square positioned to ensure that the inside portion of the test material maintained skin contact.
  Positive control: 0.4% sodium lauryl sulfate (SLS) Dose: 0.2 ml
  Negative control: Blank patch Dose: Not applicable
  Interventions: Device: Blue Non Sterile Powder Free Nitrile Examination Gloves

INTERVENTIONS:
Device: Blue Non Sterile Powder Free Nitrile Examination Gloves — Approximately 2cm x 2cm square positioned to ensure that the inside portion of the test material maintained skin contact.

SUMMARY:
Skin Sensitization Test (Modified Draize-95 Test) to Support a Low Dermatitis Potential Claim for a Blue Non Sterile Powder Free Nitrile Examination Gloves. This study is a RIPT (Repeat Insult Patch Test) to evaluate whether residual chemical additives at the level that may induce Type IV allergy in the nonsensitized general user population are present in a finished Blue Non Sterile Powder Free Nitrile Examination Glove.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be aged 18 to 65 years, inclusive;
* Subjects who have not participated in other voluntary testing for at least 30 days;
* Subjects must execute an Informed Consent Form that includes a HIPAA statement; and
* Subjects must be capable of understanding and following directions.
* Female subjects must produce a negative urine pregnancy test prior to the initiation and also at the completion of the trial.

Exclusion Criteria:

* Subjects who are in ill health, as determined by the PI;
* Subjects who are taking medication, other than birth control, which could influence the purpose, integrity or outcome of the trial;
* Subjects who have used topical or systemic corticosteroids, anti-inflammatories, antihistamines or antibiotics within 2 weeks prior to trial initiation or during their participation on this trial;
* Female subjects who are pregnant as evidenced by a urine pregnancy test, planning to become pregnant or lactating during the trial;
* Subjects who have a history of adverse reactions to cosmetics, OTC drugs, or other personal care products;
* Subjects who introduce the use of any new cosmetic, toiletry or personal care products during the trial;
* Subjects with any visible skin disease that might be confused with skin reactions caused by the test material;
* Subjects with any knowledge or indication of existing Type IV allergy (delayed hypersensitivity) to natural rubber chemical additives;
* Subjects with any indication of existing Type I allergy (immediate hypersensitivity) to natural rubber proteins;
* Subjects with a history of frequent irritation; or
* Subjects who have received endogenous or exogenous immunosuppressive treatment (or prolonged exposure to sun).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2018-06-08 (Actual)

PRIMARY OUTCOMES:
Irritation scored by Erythemal Scoring Scale | 8 weeks
  Basic Score and Description:
  0 - No visible reaction. 0.5 - Doubtful or negligible erythema reaction. 1.0 - Mild or just perceptible macular erythema reaction in a speckled/follicular, patchy or confluent pattern (slight pinking).
  2.0 - Moderate erythema reaction in a confluent pattern (definite redness). 3.0 - Strong or brisk erythema reaction that may spread beyond the test site.
  If a subject develops a positive reaction (a score value of 1.5) to the test material or shows signs of irritation after patch applications, further patching on those individuals are stopped.
  In order to qualify for the claim of a reduced sensitization potential, all 200 individuals completing the study should exhibit a score value of no more than 1.5 based on the scoring criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Caswell, Ph.D., CCRA, CCRC, Principal Investigator — Consumer Product Testing Company, Inc.
Locations (1):
- Consumer Product Testing Company, Inc., Fairfield, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No